CLINICAL TRIAL: NCT06524648
Title: A Prospective, Multicenter, Observational Pilot Study to Evaluate the Combination of niPGT-A and Morphokinetics for the Non-invasive Assessment of Embryo Development
Brief Title: International Pilot Study for Dual Non-invasive Assesment of Embryo Development
Acronym: PANDORA
Status: Recruiting | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-EES-CR-23-01
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Infertility
Keywords: Infertility; In vitro fertilization; Time lapse; niPGT-A; Embryo Development; Embryonic cell-free DNA; Morphokinetics; Artificial Intelligence; Embryo selection; Blastocyst; Ongoing pregnancy rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spent blastocyst media with embryonic cell-free DNA will be collected for DNA analysis by niPGT-A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infertile women with medical recommendation of niPGT-A: Patients will not undergo any additional intervention apart from those already scheduled for their ART. The only study specific procedures are the culture of the embryos in a timelapse system and the collection of the embryo's culture media, which is usually discarded. Both procedures will be performed following the stardard practice.
  No drugs will be administered as per the study.
  Interventions: Diagnostic Test: niPGT-A

INTERVENTIONS:
Diagnostic Test: niPGT-A — Embryos will be cultured, from oocyte fertilization up to day 6/7 of development, in a time lapse system following the standard practice. On day 6/7, embryos will be vitrified and the embryos's media will be collected for niPGT-A analysis.
  Patients will undergo a single embryo transfer (SET) following the niPGT-A report indications. In the event of 1 or more embryos with the same niPGT-A score, the embryo for transfer will be determined by the site standard practice (morphology or time-lapse score).
  Patients who do not achieve a pregnancy after a niPGT-A guided SET can undergo as many niPGT-A guided SET or COS+niPGT-A cycles as they need to get pregnant, while the study recruitment phase is active.

SUMMARY:
Choosing the best embryo is one of the major challenges for achieving success in in vitro fertilization (IVF). Traditionally, embryo evaluation has been based on morphological quality (how the embryo looks like) and chromosomal status as diagnosed by a genetic testing. However, recently new techniques that do not require manipulation of the embryo have been developed and have shown promising results.

The goal of this observational study is, by combining two non-invasive techniques, to find out some parameters during embryo development which may be related with the embryo's chromosomic status. For that, infertile women planning to undergo an IVF/ICSI treatment with a recommended niPGT-A (non-invasive Preimplantation Genetic Testing for Aneuploidies) will be invited to join the study. The main question it aims to answer is:

* Can morphokinetics parameters correlate with embryo chromosomal status?

Participants will follow their previously programmed IVF/ICSI treatment and no additional visits/interventions will be required by their participation in the study. The obtained embryos will be cultured in a time-lapse system instead of in a conventional incubator, and niPGT-A will be performed. Following the standard practice, a deferred single embryo transfer (SET) will be performed according to the niPGT-A results. After the transfer, patients will be followed-up as usual.

DETAILED DESCRIPTION:
Embryo selection represents one of the major challenges for achieving success in in vitro fertilization (IVF) cycles. Traditionally, embryo evaluation has been based on morphological quality and chromosomal status as diagnosed by a genetic testing. However, recently new non-invasive techniques that do not require additional manipulation of the embryo have been developed and have shown promising results. One such technique is the time-lapse (TL) system imaging, which considers the embryo's development in relation to its rate of division and evolution (morphokinetics). Several algorithms have been developed to aid in the selection of embryos with the highest potential for implantation by collecting data on morphokinetic events during in vitro preimplantation development. Another non-invasive method is the analysis of the cell-free desoxyribonucleic acid (cfDNA) in the culture medium, considered as a non-invasive preimplantation genetic testing for aneuploidies (niPGT-A). Despite both techniques have shown promising results, each one has its limitations, and further research is necessary to identify synergies between them with the aim of finding a more powerful approach for embryo viability evaluation.

The combination of TL and niPGT-A might have the potential to improve the embryo evaluation and thus to improve the reproductive outcome rates in IVF treatments. Therefore, the aim of the present pilot study is to identify morphokinetic parameters during embryo development in a time-lapse system which may correlate with niPGT-A results.

Once the study is approved by the competent Research Ethics Committee of each center, the recruitment and selection of patients will follow. Every potential participant will be asked to sign the study informed consent. To comply with the study design and the proposed hypothesis, an estimated total number of 200 patients will be recruited.

This is a multicenter, international, competitive, observational, prospective cohort study in which infertile women scheduled for an IVF/ICSI treatment with medical recommendation of niPGT-A will have their embryos cultured in a time-lapse system instead of in a standard incubator. On day 6/7 of embryo development, the embryo's culture medium will be collected and analyzed by niPGT-A. A subsequent embryo transfer will be performed following the niPGT-A report recommendation and participants will be followed up as routine by their gynecologist. If a pregnancy is achieved, participants will be followed up until the 12th gestational week and, if possible, until the delivery. If pregnancy is not achieved, patients can perform as many SET/COS as they need during the study recruitment period.

Data exported from the medical records and source documents will be duly codified to protect the clinical and personal information of patients in accordance with the current legislation on data protection. This information will be exported to an internal database. An interim data analysis will be carried out once the 50% of the niPGT-A cycles (100 cycles) is reached. It will help us to assess the enrollment rate, protocol compliance and an early evaluation of the study objectives.

Patient´s participation will comprise an estimated total time of up to 11 months: 1 month for the COS cycle + 1 month for the ET cycle + ≤ 9 months for the follow-up period (≤12th gestational week and ≤ 40th gestational week, when applicable).

ELIGIBILITY:
Inclusion Criteria:

* Study ICF signature.
* Female age between 20 and 42 years (bot included).
* IVF, ICSI or IVF/ICSI performed in fresh own or donated oocytes. Note: donor sperm is allowed.
* niPGT-A cases with a deferred SET (of a day 6/7 vitrified blastocyst) for any medical indication.
* Embryos cultured individually in a TL system from day 0/1 to day 6/7.

Exclusion Criteria:

* Embryos with abnormal fertilization (different from 2PN). (Note: In case of no 2PN embryos, patients may repeat the COS cycle).
* Female/couple with PGT-M and/or PGT-SR indication.
* Assisted hatching and/or artificial collapse before media collection.
* Known abnormal karyotype.
* Pathologies or malformations affecting the uterine cavity (polyps, intramural myomas ≥ 4cm or submucosal, septum or hydrosalpinx) during the patient's participation. (Note: patients are allowed to participate if the pathology is previously operated at least 3 months before patient enrollment).
* Any illness or medical condition that is unstable or which, according to medical criteria, may put at risk the patient's safety and her compliance in the study.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women complying with the selection criteria who are patients at an assisted reproduction center and, by medical recommendation, are undergoing a fertility treatment with non-invasive preimplantational genetic testing for aneuploidies.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Identification of embryo morphokinetic parameters which correlate with niPGT-A results | Up to 6/7 days
  Comparison of embryo morphokinetic parameters from the time-lapse (day 0 to day 6/7) with the niPGT-A results (informativity and ploidy)

SECONDARY OUTCOMES:
Correlation between the implantation rate (IR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | Up to 4 weeks after the embryo transfer
  Analysis to determine the correlation between morphokinetic parameters and the IR, defined as the number of gestational sacs observed by vaginal ultrasound divided by the number of embryos transferred.
Correlation between the clinical pregnancy rate (CPR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | Up to 5-6 weeks after the embryo transfer
  Analysis to determine the correlation between morphokinetic parameters and the CPR, defined as the number of pregnancies with ultrasonographic visualization of one or more gestational sacs and/or fetal heartbeat, per embryo transfer.
Correlation between the biochemical pregnancy rate (BPR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | Around 2 weeks after the embryo transfer
  Analysis to determine the correlation between morphokinetic parameters and the BPR, defined as the number of pregnancies diagnosed only by β-hCG detection (≥25 mIU/ml) without a gestational sac visualized by vaginal ultrasound, per number of pregnancies.
Correlation between the ectopic pregnancy rate (EPR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | Up to 4-5 weeks after the embryo transfer
  Analysis to determine the correlation between morphokinetic parameters and EPR, defined as the number of pregnancies outside the uterine cavity, diagnosed clinically, hormonally, by ultrasound, surgical visualization or histopathology, per number of pregnancies.
Correlation between the clinical miscarriage rate (CMR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | Over 12 gestational weeks
  Analysis to determine the correlation between morphokinetic parameters and the CMR, defined as the number of spontaneous pregnancy losses before the 12th gestational week, in which a gestational sac/s was previously observed and heartbeat detected, per number of pregnancies.
Correlation between the ongoing pregnancy rate (OPR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | ≥12 gestational weeks
  Analysis to determine the correlation between morphokinetic parameters and the OPR, defined as the number of pregnancies of, at least,12 gestational weeks (at least one fetus with a discernible heartbeat diagnosed) achieved per each embryo transfer.
Correlation between the Live Birth Rate (LBR) and embryo morphokinetic parameters in the niPGT-A guided single embryo transfer (SET) | 40 gestational weeks
  Analysis to determine the correlation between morphokinetic parameters and the LBR, defined as the number of live births per embryo transfer. Live birth is defined as the complete expulsion or extraction from a woman of a product of conception after 22 weeks of gestation, which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.
Identification of morphokinetic parameters which might predict the optimal time for media collection. | Up to 6/7 days of embryo development
  Comparison of niPGT-A informativity results with morphokinetic parameters
To explore the relationship between niPGT-A results and morphokinetics with the type of ovarian stimulation and induction, the patient's intertility history and embryo quality | Over 3-4 weeks
  Multivariant analysis to determine how the relationship between niPGT-A results and morphokinetics is affected by ART/patient variables: type of ovarian stimulation and induction, the patient's intertility history (previous miscarriages, known infertility causes, previous implantation failures), and embryo quality (determined by standard morphology evaluation).
Identification of the correlation between morphokinetic parameters and spent blastocyst media contamination | Up to 6/7 days of embryo development
  Correlate morphokinetic parameters with the presence of maternal and/or external DNA in the culture media for niPGT-A
Comparison of the products of conception (POC) results with the niPGT-A results | Up to 12 gestational weeks
  Correlate the niPGT-A results with the POC results
To study the relathionship among the morphokinetics, niPGT-A and the patient's body mass index (BMI) | Up to 6/7 days
  To anlyse the patient's BMI influence on the correlation between morphokinetics and niPGT-A, only when own oocytes are used.

OTHER OUTCOMES:
To evaluate the relathionship of the cell-free DNA (cfDNA) concentration of the spent blastocyst media (SBM) with morphokinetic parameters and/or niPGT-A | Up to 6/7 days of embryo development
  To assess the cfDNA concentration in a 20% of the SBMs and evaluate its correlation with morphokinetic parameters and/or niPGT-A

CONTACTS AND LOCATIONS:
Overall Officials: Luis Navarro, PhD, Principal Investigator — Igenomix; Carmen Rubio, PhD, Study Chair — Igenomix
Locations (8):
- Kinderwunsch Institut Schenk, Dobl, Austria
- Spain (6):
  - Fertty, Barcelona, Barcelona
  - Hospital Ruber Internacional, Madrid, Madrid
  - Next Fertility Murcia, Murcia, Murcia
  - Next Fertility Sevilla, Seville, Sevilla
  - Next Fertility Valencia, Valencia, Valencia
  - Vida Recoletas Sevilla, Seville
- Orchid IVF Clinic, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No